CLINICAL TRIAL: NCT03524911
Title: Choose Health: Food, Fun, and Fitness Curriculum Promotes Positive Behaviors in 3rd-5th Graders Compared to Control Period
Brief Title: Choose Health: Food, Fun, and Fitness Curriculum Promotes Positive Behaviors in 3rd-5th Graders Compared to Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHFFF0518
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Childhood Obesity; Nutrition Poor
Keywords: Nutrition education; Evaluation; Child diet; EFNEP
MeSH Terms: conditions — Pediatric Obesity; Malnutrition

STUDY DESIGN:
Intervention Model Description: Delayed intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHFFF nutrition education (Experimental): Expanded Food and Nutrition Education (EFNEP) participants in 5 NY counties in 2015
  Interventions: Behavioral: CHFFF nutrition education

INTERVENTIONS:
Behavioral: CHFFF nutrition education

SUMMARY:
The Choose Health: Food, Fun, and Fitness (CHFFF) curriculum was evaluated in 3rd-5th graders, hypothesizing that change pre- to post- CHFFF education would be greater than in the same child during a delayed intervention control period.

DETAILED DESCRIPTION:
Choose Health: Food, Fun, and Fitness (CHFFF) is a Cornell curriculum for 3rd-6th graders targeting behaviors to prevent obesity and chronic disease risk: fewer sweetened drinks; more vegetables, fruits, and whole grains; fewer high-fat and high-sugar foods; and active play. The 6 lessons use experiential learning, food preparation, active games, goal setting, and a family newsletter. It was evaluated in 561 Expanded Food and Nutrition Education (EFNEP) participants in 27 after-school and 28 in-school groups in 5 NY counties in 2015 using a quasi-experimental design, with a delayed-intervention control period prior to CHFFF. Youth completed a self-reported survey 3 times: at initial enrollment, after a 6-week no-intervention control period, and after receiving the 6 weekly CHFFF lessons. Outcome measures included dietary intake scores created based on factor analysis, and related precursors. It was hypothesized that change pre- to post- CHFFF education would be greater than in the same child during the delayed intervention control period. Following CHFFF, youth improved significantly (p<.05) compared to their control period in overall diet quality, vegetable intake, fruit intake, soda/fast food intake and choice, and the frequency with which they read nutrition facts labels, shared about healthy eating with their family, and tried a new food.

ELIGIBILITY:
Inclusion Criteria:

* Participants in EFNEP nutrition education in schools and in after-school programs in 5 counties in NY during the 2014-2015 school year

Exclusion Criteria:

* Younger than 3rd grade (n=3)
* Those with fewer than 4 lessons (n=9)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 561 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2015-06-11 (Actual); Study Completion 2015-06-11 (Actual)

PRIMARY OUTCOMES:
Child Diet | Youth completed the survey at initial enrollment, after a 6-week delayed-intervention control period, and after receiving CHFFF.
  Dietary intake was assessed via a self-reported survey, then 4 dietary scores were created based on factor analysis: overall diet quality, vegetable intake, fruit intake, and soda/fast food intake.

SECONDARY OUTCOMES:
Psychosocial mediators | Youth completed the survey at initial enrollment, after a 6-week delayed-intervention control period, and after receiving CHFFF.
  Assessed via a self-report survey, these included soda/fast food choices, and the frequency with which they read nutrition facts labels, shared about healthy eating with their family, and tried a new food.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Wolfe, PhD, Principal Investigator — Cornell University Division of Nutritional Sciences

IPD SHARING:
Plan to Share IPD: Yes
Submitting all collected IPD to the Ag Data Commons at the USDA National Agricultural Library.
Time Frame: Plan to submit in May 2018
Access Criteria: Public access
URL: https://data.nal.usda.gov/about-ag-data-commons

REFERENCES:
- See also: Choose Health: Food, Fun, and Fitness curriculum and related resources — http://fnec.cornell.edu/for-partners/curricula/chfff/